CLINICAL TRIAL: NCT06487481
Title: A Phase I Dose-escalation Study of Preoperative Radiation Therapy in Participants With Resectable Recurrent Abdominal Adrenocortical Carcinoma
Brief Title: Study of Preoperative Radiation Therapy in Participants With Resectable Recurrent Abdominal Adrenocortical Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001587; 001587-C
Record Dates: First submitted 2024-07-03; First posted 2024-07-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-08

CONDITIONS: Adrenocortical Carcinoma (ACC); Recurrent Adrenocortical Carcinoma (ACC); Recurrent Abdominal Adrenocortical Carcinoma (ACC); Carcinoma, Adrenocortical; Carcinoma, Adrenal Cortical
Keywords: external beam radiation therapy (EBRT); abdominal adrenocortical carcinoma (ACC); preoperative radiation; Mitotane; Maximum Tolerated Dose (MTD); Surgical Resection; in-field intraabdominal progression-free survival (PFS); out-of-field intraabdominal progression-free survival (PFS); DNA damage repair markers; oxidative stress response
MeSH Terms: conditions — Adrenocortical Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preop RT + surgery (Experimental): Preoperative RT at escalating doses followed by surgical resection
  Interventions: Procedure: Surgical resection; Radiation: Preoperative RT

INTERVENTIONS:
Procedure: Surgical resection — Planned surgical resection (all participants) 4 weeks after completion of the preoperative RT
Radiation: Preoperative RT — Preoperative RT at escalating doses in daily fractions over approximately 2-3 weeks; 2 weeks (DL1), or 3 weeks (DL2 or DL3) based on assigned Cohort and Dose Level (DL). Cohorts are by mitotane status at enrollment: Cohort 1 (with detectable mitotane levels), Cohort 2 (never had or without detectable mitotane levels), Cohort 3 (either).

SUMMARY:
Background:

Adrenocortical carcinoma (ACC) is a rare cancer of the adrenal glands. ACC often returns after tumors are removed with surgery. Less than 35% of people with ACC survive 5 years after diagnosis.

Objective:

To test a new type of external beam RT before surgery in people with ACC.

Eligibility:

People aged 18 years and older with ACC that came back after treatment but may be safely removed with surgery.

Design:

Participants will be screened. They will have a physical exam with blood and urine tests. They will have tests of their heart function. They will have imaging scans. A small sample of tumor tissue may be collected if one is not available. They will undergo laparoscopy: Small incisions will be made in the abdomen so that a thin tube with a light and camera can be inserted to view the organs.

RT comes from a machine that aims radiation at tumors. Participants will receive preoperative RT in daily fractions over approximately 2-3 weeks, followed by a planned surgical resection about 4 weeks after the completion of RT. Visits will last 30 to 60 minutes.

Participants will undergo surgery to remove their tumors about 4 weeks after they finish RT. They will stay in the hospital 1 to 3 weeks after surgery.

Participants will have follow-up visits for 10 years after surgery.

DETAILED DESCRIPTION:
Background:

* Although surgical resection is the treatment of choice in participants with localized or regionalized primary and recurrent abdominal adrenocortical carcinoma (ACC), loco-regional recurrence following complete resection of ACC occurs in 50-80% of the participants, most commonly in the first five years postoperatively.
* Retrospective single institutional series report improvement in local control with postoperative adjuvant radiotherapy (RT) in selected participants with ACC.
* Preoperative RT is used in several abdominal and retroperitoneal malignancies to improve local control. There is no prospective data available for the use of this treatment approach for participants with resectable ACC.
* We hypothesize that preoperative RT alone is safe and can result in a lower loco-regional recurrence in participants with resectable recurrent ACC with no peritoneal carcinomatosis. Thus, this phase I dose-escalation trial aims to evaluate the safety and feasibility of preoperative RT in participants with resectable recurrent ACC.
* Health-related quality of life (QOL) is a well-accepted tool to measure the outcome of cancer treatments. SF-36 V1 questionnaire has been frequently used to evaluate the QOL in participants with cancer. There is no study evaluating the difference in QOL in participants with resectable recurrent ACC undergoing preoperative RT and surgery.

Objectives:

-To determine the maximum tolerated dose and the safety and toxicity profile of preoperative external beam RT with or without standard of care mitotane, before surgical resection in participants with resectable ACC

Eligibility:

* Age >= 18 years
* Pathological confirmation of ACC with clinical evidence of abdominal recurrence
* ECOG 0-2
* Surgically resectable disease at presentation with no or limited extra-abdominal disease and without ACC peritoneal carcinomatosis based on a diagnostic laparoscopy at screening.
* The last dose of chemotherapy treatment except for mitotane more than 4 weeks prior to starting treatment with this protocol, and participants must have recovered from chemotherapy.
* No prior abdominal RT
* No contraindication to abdominal RT

Design:

* This study will enroll up to 24 evaluable participants as follows:

  * Participants will be enrolled in Cohort 1 or 2 based on mitotane use or serum level. Up to 6-18 evaluable participants per these cohorts (i.e., resectable ACC with and without mitotane use) will be enrolled to assess the safety of 3-level dose-escalating preoperative RT.
  * Participants will be enrolled in Cohort 3 regardless of mitotane use or serum level, and will only start enrollment when we observe no DLTs in > 1 participant in Cohort 1 at Dose Level 1. Up to 12 evaluable participants will be enrolled in this cohort.
* Preoperative assessment of QOL using a standardized questionnaire (SF-36 V1) will be obtained at baseline.
* Participants will be treated with preoperative RT, followed by a planned surgical resection, 4 weeks after the completion of RT.
* A standard "3 + 3" design will be used to determine the MTD of dose-escalated RT, with 3 dose levels (DL1- 30 Gy delivered in 10 fractions, DL2-36 Gy in 12 fractions, DL3-42 Gy in 14 fractions).
* Postoperative surveillance imaging studies and laboratory tests will be performed every 3 months in the first 3 years, then every 6 months thereafter in years 4-10. FDG-PET scan will be performed every 6 months postoperatively in the first 3 years, then every year in years 4-10. Additional assessments may be performed if clinically indicated.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age >= 18 years
* Pathological confirmation of ACC by the Laboratory of Pathology, NCI. Note: Confirmation may be done from archival sample; fresh tissue is not required unless otherwise acquired for clinical purposes.
* Measurable disease by RECISTv1.1. criteria at enrollment
* Evidence of recurrent ACC amenable to surgical resection that can be performed at NIH Clinical Center (CC)
* Must be suitable for external beam radiotherapy AND surgery in the opinion of the treating investigator (e.g., based on clinical history and imaging)
* Participants with metastatic ACC outside the area(s) to be exposed to investigational treatments (e.g., liver parenchyma, lung[s], or bone[s]) must have disease that is amendable for a complete resection and/or catheter-based and/or radiation-based ablation.
* Mitotane therapy- Participants may be receiving mitotane currently, have received it in the past, or never have received mitotane. However, participants will be evaluated in separate cohorts based on mitotane use and, as enrollment is sequential, not all participants may be eligible for the study at all times. Note: Participants with a history of mitotane use may continue on study at the discretion of the treating investigator. Participants will not initiate mitotane on study.
* Participants must agree to undergo tumor biopsy of easily accessible tumor sites prior to study treatment.
* Performance Status (ECOG) 0-2
* Adequate organ function, including:

  * Hemoglobin >= 9.0 gm/dL
  * ANC >= 1,500/mm^3
  * Platelets >= 75,000/mm^3
  * AST and ALT <= 3 x Upper Limit Normal (ULN)
  * Bilirubin <= 2 x ULN
  * Creatinine within normal institutional limits or creatinine clearance >60 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal calculated using eGFR.
* Individuals of childbearing potential must agree to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) prior to RT and continue until at least 4 months following cytoreduction surgery.
* Nursing (including breastfeeding) participants must agree to discontinue nursing prior to RT and continue until at least 4 months following cytoreductive surgery.
* Ability of participant to understand and willingness to sign a written informed consent document
* Participants must agree to co-enroll in tissue collection protocol 09C0242 "Prospective comprehensive molecular analysis of endocrine neoplasms."

EXCLUSION CRITERIA:

* Primary ACC or suspicious/indeterminate adrenal tumor without pathological confirmation
* Prior abdominal radiation therapy
* Participants who have received chemotherapy, immunotherapy, investigational therapy, or radiotherapy treatment within the last 4 weeks prior to starting treatment and/or have not recovered from toxicities to less than grade 2 CTCAE.
* Infection requiring parenteral antibiotics
* Suspected or proven ACC peritoneal metastasis
* Pre-existing known or suspected radiation sensitivity syndromes
* Prohibitive condition(s) to diagnostic laparoscopy
* Participants who have an unacceptable risk for a major surgical procedure such as participants with high risks for major cerebro-cardiovascular (such as those who had doxorubicin exposure as based on screening echocardiogram and ECG) and pulmonary complications and those with estimated perioperative mortality greater than 15% per ACS NSQIP Surgical Risk calculator.
* Participants receiving other investigational therapies
* Participant pregnancy
* Active systemic infections, coagulation disorders, or other major medical illnesses such as uncontrolled diabetes mellitus, uncontrolled hypertension (persistently grade 2 or worse), active severe cerebro-cardio-pulmonary diseases, and acute major organ dysfunction.
* Acute intraabdominal conditions such as obstruction or peritonitis at the time of the evaluation or surgery.
* Evidence at screening of or currently active CNS metastasis within 6 months of RT; participants with history of treated brain metastases with intracranial recurrence within 6 months prior to treatment. Note: Participants with any signs or symptoms suggestive of previously undiagnosed brain metastasis at screening or with a history of brain metastasis should receive imaging at screening; otherwise, imaging is not required.
* HIV-positive participants with CD4 below 200 or who are not on anti-retroviral therapy
* Participants who have a history of another primary malignancy from which the participant has been disease-free for < 3 years at the time of enrollment.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2030-12-01 (Estimated); Study Completion 2040-12-01 (Estimated)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) and safety and toxicity profile of preoperative external beam radiation therapy (RT) with or without standard-of-care mitotane, before surgical resection in participants with resectable recurrent ACC | from the start of RT and for 30 days after its completion
  Fraction of participants with a dose-limiting toxicity (DLT) will be reported at each dose level

SECONDARY OUTCOMES:
Determine the 30-day postoperative complications per Clavien-Dindo classification | baseline, until 30 days after cytoreductive surgery
  Assessment of 30-day postoperative RT complications determined by Clavien-Dindo classification (frequency and and severity)
Determine the objective response of ACC within the radiation treatment field per RECIST criteria | baseline, every 3-6 months after cytoreductive surgery for up to 10 years after surgery
  Objective response determined by RECIST, results as fraction in evaluable participants and by 95% confidence interval of the median
Assess in-field intraabdominal progression-free survival (PFS) | baseline, every 3-6 months after cytoreductive surgery for up to 10 years after surgery
  In-field intraabdominal progression-free survival (PFS) determined by RECIST using the Kaplan-Meier method and by 95% confidence interval of the median
Determine overall survival (OS) through 10 years postoperatively | baseline, every 3-6 months after cytoreductive surgery for up to 10 years after surgery
  Overall survival (OS) up to 10 years postoperatively determined by RECIST using the Kaplan-Meier method and by 95% confidence interval of the median
Assess quality of life measured by Short Form-36 Health Survey version 1.0 (SF-36 V1) questionnaire | baseline, 4 weeks after RT, and then 2 weeks, 4 weeks, 6 months and 12 months after surgery
  Quality of life (QOL) measured by SF-36 V1 questionnaire evaluated using appropriate paired tests and descriptive results

CONTACTS AND LOCATIONS:
Overall Officials: Naris Nilubol, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded will be shared upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested from other researchers within 10 years after the completion of the primary endpoint by contacting the Principal Investigator.
Access Criteria: Data from this study may be requested by contacting the PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001587-C.html